CLINICAL TRIAL: NCT03430791
Title: A Phase I/II Trial of Combination Tumor Treating Fields, Nivolumab Plus/Minus Ipilimumab for Recurrent Glioblastoma
Brief Title: Trial of Combination Tumor Treating Fields (TTF; Optune), Nivolumab Plus/Minus Ipilimumab for Recurrent Glioblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study Investigator/Sponsor decided to end enrollment earlier.
Sponsor: Baptist Health South Florida (Other)
Collaborators: Bristol-Myers Squibb (Industry); NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-ODI-002
Record Dates: First submitted 2018-01-31; First posted 2018-02-13 (Actual); Results first posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2022-11

CONDITIONS: Recurrent Glioblastoma
Keywords: recurrent glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: This is an open-label, phase II trial with two parallel arms, two-stage design and appropriate stopping rules for poor efficacy. Arm A will enroll participants without prior PD1/PDL1 checkpoint inhibitor, while Arm B will enroll participants with prior PD1/PDL1 checkpoint inhibitor. The investigator expect to enroll at least 30 (15 in each Arm) and a maximum of 60 (30 in each Arm) evaluable subjects. All subjects will receive tumor treating field (TTF) therapy plus nivolumab infusions for a maximum of 24 months, plus/minus concurrent ipilimumab for a maximum of 4 doses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Nivolumab Monotherapy (Experimental): Nivolumab 240 mg IV every 2 weeks for maximum of 24 months. TTF (Optune) for max of 24 months
  Interventions: Drug: Nivolumab 240 mg IV; Device: NovoTTF200A (Optune)
- Nivolumab+Ipilimumab (Experimental): Nivolumab 3 mg/kg IV with ipilimumab then 240 mg every 2 weeks for maximum of 24 months.
  Ipilimumab 1 mg/kg IV every 6 weeks maximum of 4 times. NovoTTF200A (Optune) TTF for maximum 24 months
  Interventions: Drug: Nivolumab 240 mg IV; Drug: Nivolumab 3 mg/kg; Drug: Ipilimumab 1 mg/kg; Device: NovoTTF200A (Optune)

INTERVENTIONS:
Drug: Nivolumab 240 mg IV — Nivolumab IV 240mg IV every 2 weeks for maximum of 24 months.
  Other Names: Nivolumab Monotherapy
Drug: Nivolumab 3 mg/kg — Nivolumab IV 3mg/kg every 2 weeks for maximum of 24 months.
  Other Names: Nivolumab+Ipilimumab
  Arms: Nivolumab+Ipilimumab
Drug: Ipilimumab 1 mg/kg — Ipilimumab IV 1 mg/kg every 6 weeks for maximum of 4 doses.
  Other Names: Nivolumab+Ipilimumab
  Arms: Nivolumab+Ipilimumab
Device: NovoTTF200A (Optune) — A device to be worn continuously for a goal of 75% of the time, ranging from 18 hours daily nonstop or 22 hours daily with 2-3 days off monthly.

SUMMARY:
Phase I/II trial in which participants with recurrent glioblastoma will receive a combination of tumor treating fields(portable device), nivolumab with or without ipilimumab.

DETAILED DESCRIPTION:
Phase I/II trial in which participants with recurrent glioblastoma will receive a combination of tumor treating fields(portable device), nivolumab with or without ipilimumab.

The NovoTTF200A (OptuneTM) device is worn continuously for a goal of 75% or more of the time, ranging from at least 18 hours daily uninterrupted or 22 hours daily with 2-3 days off monthly. Therapy is planned for approximately 24 months.

Infusions with nivolumab will start within 1 week of study start. Ipilimumab will either start with the second nivolumab infusion or at after tumor progression. Nivolumab is infused intravenously at 240 mg once every 2 weeks with or without ipilimumab for a maximum of 24 months. Ipilimumab is dosed at 1 mg/kg once every 6 weeks for a maximum of 4 doses (24 weeks). Infusions will continue until maximum doses are completed or there is confirmed tumor progression, intolerable adverse effects or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed World Health Organization Grade IV glioblastoma with supratentorial distribution.
* Unequivocal evidence of progressive disease on contrast-enhanced brain CT or MRI as defined by Response Assessment in Neuro-Oncology (RANO) criteria, or documented recurrent glioblastoma on biopsy.
* Measurable disease based on RANO criteria.
* Prior therapies including radiation and temozolomide.
* Any number of recurrences are allowed. Resection of recurrent glioblastoma is not considered a prior treatment.
* From the projected start date of study treatment, the following periods must have elapsed: 4 weeks from any investigational agent, 4 weeks from cytotoxic therapy (except 23 days for temozolomide and 6 weeks from nitrosoureas), or 4 weeks from any other antibodies or any other antineoplastic therapies.
* Must be at least 12 weeks from radiotherapy or progression outside of the high-dose radiation target volume or unequivocal evidence of progressive tumor on biopsy.
* All adverse events Grade > 1 related to prior therapies (chemotherapy, radiotherapy, and/or surgery) must be resolved, except for alopecia.
* Karnofsky Performance Status (KPS) ≥ 60
* Adequate organ and marrow function as defined below, all screening labs should be performed within 14 days of treatment initiation:

  * absolute neutrophil count ≥ 1,000/mcL
  * platelets ≥100,000/mcL
  * hemoglobin > 8.0 mg/dL
  * total bilirubin ≤ 2.0 x upper limit of normal
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 × upper limit of normal
  * creatinine or creatinine clearance ≥ 60 mL/min/1.73 m2 for creatinine >ULN
* Corticosteroid dose must be stable or decreasing for at least 5 days prior to enrollment.
* Nivolumab and ipilimumab are potentially teratogenic or abortifacient. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to entry and for the duration of study. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Male subjects should agree to use adequate method of contraception starting with the first dose through 7 months after the last dose of therapy.
* Brain CT or MRI within 14 days prior to start of study drug.
* Archival tissue for evaluation of correlative objectives (if available).
* Ability to understand and the willingness to provide written informed consent.

Exclusion Criteria:

* Infratentorial disease.
* Bevacizumab within 2 months of enrollment. Prior use of ipilimumab or other CTLA-4 inhibitor or prior TTFields.
* Tumors with known IDH1 (isocitrate dehydrogenase 1) or IDH2 mutations as determined by immunohistochemistry for the IDH1 R132H variant or by direct sequencing. IDH1/2-mutant gliomas have a prolonged overall survival rate compared to IDH1/2-wildtype gliomas, indicating distinct natural history.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab or ipilimumab or their excipients.
* Current or planned participation in a study of an investigational agent or using an investigational device.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Active or life-threatening infection requiring intravenous or >2 weeks of systemic therapy.
* Prior stereotactic radiotherapy, convection enhanced delivery (CED) or brachytherapy requires a biopsy to confirm radiographic progression is consistent with progressive tumor and not treatment-related necrosis unless the recurrent lesion is outside of any prior high-dose radiation target volume or distant from the prior CED or brachytherapy site.
* There is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, so breastfeeding must be discontinued by enrollment on study.
* Uncontrolled HIV or AIDS is not allowed. Patients with known history of HIV but with undetectable viral load on antiretroviral therapy are allowed.
* Congestive heart failure, myocardial infarction, or hemorrhagic/ischemic stroke in the last 3 months.
* Active illicit drug use or diagnosis of alcoholism
* Known additional malignancy that is progressing or requires active treatment within 3 years of start of study drug. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer or other in situ malignancy that has undergone potentially curative therapy and/or with >90% probability of survival beyond 5 years.
* Any surgery (not including minor diagnostic procedures such as lymph node biopsy) within 2 weeks of start of treatment. Incomplete recovery from any side effects of previous procedures is also exclusionary.
* Any significant autoimmune disorders expected to impact multiple or internal organs, excluding mild eczema or autoimmune thyroiditis treated with thyroidectomy and requiring systemic immunosuppressive or immunomodulatory therapy.
* Any implanted programmable cranial device, including reprogrammable ventriculoperitoneal shunt (VPS) or cochlear implants, that precludes use of TTFields (Optune) therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2021-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yazmin Odia, Principal Investigator — Miami Cancer Institute at Baptist Health, Inc.
Locations (1):
- Miami Cancer Institute at Baptist Health, Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Miami Cancer Institute website — http://baptisthealth.net/cancer-care/home

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab+Ipilimumab: Nivolumab 3 mg/kg IV with ipilimumab then 240 mg every 2 weeks for maximum of 24 months.
  Ipilimumab 1 mg/kg IV every 6 weeks maximum of 4 times. NovoTTF200A (Optune) TTF for maximum 24 months
  Nivolumab 240 mg IV: Nivolumab IV 240mg IV every 2 weeks for maximum of 24 months.
  Nivolumab 3 mg/kg: Nivolumab IV 3mg/kg every 2 weeks for maximum of 24 months.
  Ipilimumab 1 mg/kg: Ipilimumab IV 1 mg/kg every 6 weeks for maximum of 4 doses.
  NovoTTF200A (Optune): A device to be worn continuously for a goal of 75% of the time, ranging from 18 hours daily nonstop or 22 hours daily with 2-3 days off monthly.
Period: Overall Study
Arm/Group | Nivolumab Monotherapy | Nivolumab+Ipilimumab
Started | 4 | 0
Completed | 4 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants with prior PD1/PDL1 checkpoint inhibitor were enrolled, thus no participants were assigned to the Nivolumab+Ipilimumab arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab Monotherapy | Nivolumab+Ipilimumab | Total
Number analyzed (Participants) | 4 | 0 | 4
Age, Continuous [Median (Full Range); unit: Years] | 65 [57 to 80] |  | 65 [57 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 0 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate According to Modified iRANO Criteria
Description: Objective response rate is the proportion of patients whose best overall response per modified immunotherapy response assessment in neuro-oncology (iRANO) criteria is complete (CR) or partial (PR) after at least 6 weeks from start of therapy
Time Frame: 2 years
Population: No participants met criteria for the Nivolumab+Ipilimumab arm, thus none were enrolled in that arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab Monotherapy | Nivolumab+Ipilimumab
Number analyzed (Participants) | 4 | 0
Participants | 0 |

2. Secondary Outcome: Objective Response Rate (ORR) by Standard RANO Criteria
Description: Objective response rate is the proportion of patients whose best overall response per response assessment in neuro-oncology (RANO) criteria is complete (CR) or partial (PR) after at least 6 weeks from start of therapy
Time Frame: 2 years
Population: No participants met criteria for the Nivolumab+Ipilimumab arm, thus none were enrolled in that arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab Monotherapy | Nivolumab+Ipilimumab
Number analyzed (Participants) | 4 | 0
Participants | 0 |

3. Secondary Outcome: Progression Free Survival (PFS)
Description: The length of time that a participant lives with the disease but it does not get worse.
Time Frame: 2 years
Population: No participants met criteria for the Nivolumab+Ipilimumab arm, thus none were enrolled in that arm.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nivolumab Monotherapy | Nivolumab+Ipilimumab
Number analyzed (Participants) | 4 | 0
days | 62.5 (16.1) |

4. Secondary Outcome: Number of Toxicities
Description: Total number of toxicities as defined by AEs that attributed as probable or possibly related to the study drug across all study subjects.
Time Frame: Up to 2 years
Population: No participants met criteria for the Nivolumab+Ipilimumab arm, thus none were enrolled in that arm.
Measure: Number; unit: adverse events
Arm/Group | Nivolumab Monotherapy | Nivolumab+Ipilimumab
Number analyzed (Participants) | 4 | 0
adverse events | 13 |

5. Secondary Outcome: Rate of Treatment Compliance
Description: Percent of participants who have a compliance rate above the 75% goal for tumor treating fields (TTFields) therapy via the NovoTTF200A (OptuneTM). Daily compliance rates for using the device are averaged (mean ± stdev) over the 28-31 days of the month.
Time Frame: Monthly for up to 2 years
Population: No participants met criteria for the Nivolumab+Ipilimumab arm, thus none were enrolled in that arm.
Measure: Mean (Standard Deviation); unit: percent of participants compliant
Arm/Group | Nivolumab Monotherapy | Nivolumab+Ipilimumab
Number analyzed (Participants) | 4 | 0
percent of participants compliant | 75 (12) |

6. Secondary Outcome: Discontinuation Rate of Any Component of Therapy
Description: Proportion of participants who discontinued therapy. Reasons for discontinuation also will be noted.
Time Frame: Up to 2 years
Population: No participants met criteria for the Nivolumab+Ipilimumab arm, thus none were enrolled in that arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab Monotherapy | Nivolumab+Ipilimumab
Number analyzed (Participants) | 4 | 0
Participants | 4 |

7. Secondary Outcome: Change in Quality of Life From Baseline Using the Functional Assessment of Cancer Therapy-Brain (FACT-Br)
Description: FACT-Br is a validated self-report tool measuring general quality of life (QOL) that assesses symptoms or problems associated with CNS tumors across 5 scales. FACT-Br yields data about total QOL, as well as dimensions of disease specific physical, social/family, emotional, and functional well-being. The tool contains 20 items using a 5-point Likert scale. A higher score indicates better QOL, ranging from 0 (lowest) to 92 (highest). Median percent change between first and last measurement provided, with negative percent change indicating a decline in function.
Time Frame: Up to 2 years
Population: No participants met criteria for the Nivolumab+Ipilimumab arm, thus none were enrolled in that arm.
Measure: Median (Full Range); unit: percentage of change
Arm/Group | Nivolumab Monotherapy | Nivolumab+Ipilimumab
Number analyzed (Participants) | 4 | 0
percentage of change | -22 [-25 to 3] |

8. Secondary Outcome: Change in Quality of Life From Baseline Using the Functional Assessment of Cancer Therapy-General (FACT-G)
Description: FACT-G is a validated self-report tool measuring general quality of life (QOL) that assesses symptoms or problems associated with any tumors. The tool contains 33 items using a 5-point Likert scale. A higher score indicates better QOL, ranging from 0 (lowest) to 108 (highest). Median percent change between first and last measurement provided, with negative percent change indicating a decline in function.
Time Frame: Up to 2 years
Population: No participants met criteria for the Nivolumab+Ipilimumab arm, thus none were enrolled in that arm.
Measure: Median (Full Range); unit: percentage of change
Arm/Group | Nivolumab Monotherapy | Nivolumab+Ipilimumab
Number analyzed (Participants) | 4 | 0
percentage of change | -13 [-28 to 3] |

ADVERSE EVENTS:
Time Frame: 18 months
Description: No participants were accrued to the Nivolumab+Ipilimumab arm, thus the number at risk for SAE, all-cause mortality, and other events is 0 for that arm.
Arm/Group | Nivolumab Monotherapy | Nivolumab+Ipilimumab
All-Cause Mortality (participants affected / at risk) | 2/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 4/4 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab Monotherapy (N=4) | Nivolumab+Ipilimumab (N=0)
Fatigue (General disorders) | 1 (2) | 0
Scalp rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0
Dry mouth (Gastrointestinal disorders) | 1 (1) | NA
Dysarthria (Nervous system disorders) | 1 (1) | NA
Fall (Injury, poisoning and procedural complications) | 1 (1) | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | NA
Hemiplegia (Nervous system disorders) | 1 (1) | NA
Hyperthyroid (Endocrine disorders) | 1 (1) | NA
Pituitary disorder (Endocrine disorders) | 1 (1) | NA
Seizure (Nervous system disorders) | 1 (1) | NA
Stomach pain (Gastrointestinal disorders) | 1 (3) | NA
Toenail avulsion (Skin and subcutaneous tissue disorders) | 1 (1) | NA
Weakness (General disorders) | 2 (2) | NA
Urinary tract infection (Infections and infestations) | 1 (1) | NA
Worsening herpes zoster infection (Infections and infestations) | 1 (1) | NA

LIMITATIONS AND CAVEATS:
Did not accrue the target number of participants needed to achieve target power and statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT03430791/Prot_SAP_001.pdf